CLINICAL TRIAL: NCT05659095
Title: A Randomized-controlled Clinical Trial to Treat Chinese Advanced AGA With Autologous Hair Follicle Derived Mesenchymal Stem Cell Suspension
Brief Title: Autologous Hair Follicle Derived Mesenchymal Stem Cell Suspension to Treat AGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: NFEC-2020-245
Record Dates: First submitted 2022-10-10; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-10

CONDITIONS: Hair Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment groups (Experimental): Healthy hair follicles were extracted from the occipital area and treated to obtain hair follicle mesenchymal stem cells suspensions. The recipient sites were divided into two groups. Nine points were injected in a 1 cm2 area, and 100 μl of solution containing either 1 × 105 cells or normal saline was injected at each point.
  Interventions: Other: autologous hair follicle derived mesenchymal stem cell suspension
- Control groups (No Intervention): The control group was injected with the same volume of normal saline.

INTERVENTIONS:
Other: autologous hair follicle derived mesenchymal stem cell suspension — Healthy hair follicles were extracted from the occipital area and treated to obtain hair follicle mesenchymal stem cells suspensions. The recipient sites were divided into two groups. Nine points were injected in a 1 cm2 area, and 100 μl of solution containing either 1 × 105 cells or normal saline was injected at each point. The follow-up duration was 9 months.
  Arms: Experiment groups

SUMMARY:
Androgenic alopecia (AGA) is characterized by progressive hair follicle miniaturization, and novel treatments are needed to intervene in the miniaturization process. The investigators aimed to evaluate the efficacy, safety, effectiveness, and effective population of autologous hair follicle mesenchymal stem cell therapy for the treatment of advanced AGA in Chinese people.

50 participants ranging from 25 to 45 years old, with an average age of 32 ± 1.24 years were included. None of them had ever used minoxidil, finasteride, or other drugs to promote hair growth. Healthy hair follicles were extracted from the occipital area and treated to obtain hair follicle mesenchymal stem cells suspensions. The recipient sites were divided into two groups. Nine points were injected in a 1 cm2 area, and 100 μl of solution containing either 1 × 105 cells or normal saline was injected at each point. The follow-up duration was 9 months. Observers were blinded to patient groupings and measurements.

DETAILED DESCRIPTION:
Androgenic alopecia (AGA) is the most common form of hair loss. It starts in adolescence and is mainly characterized by progressive hair follicle miniaturization. In the continuous hair cycle process, the pathological hair follicle mesenchymal niche in the hair loss area is continuously damaged. The mesenchymal cells are continuously consumed, resulting in functional disorder, gradually losing the ability to induce the proliferation and differentiation of hair follicle epidermal cells to form hair follicles. This process eventually leads to the complete miniaturization and loss of hair follicles. Presently, non-surgical treatments for AGA, such as minoxidil or finasteride, have great individual differences in the effectiveness in different populations and may not achieve the expected effect of patients with advanced AGA, although they are still recommended as first-line drugs for androgenic alopecia.

Hair follicle mesenchymal stem cells (HF-MSCs) included dermal papilla cells (DPCs) and dermal sheath cells (DSCs). Similar to other types of mesenchymal stem cells, HF-MSCs possess stem cell characteristics such as multidirectional differentiation potential, the ability of integrated homing to a specific niche, and secretion of exosomes and cytokines, which have great application prospects. HF-MSCs are considered an important therapeutic agent to promote hair growth. A previous study has indicated that injection of DPC spheres can promote hair growth on the back of mice. A double-blind clinical trial in Japan confirmed that treatment of the expanded dermal sheath cup cells (DSCCs) of healthy human hair follicles could promote the growth of hair follicles in the hair loss area of the forehead. However, the population and stage of AGA for which HF-MSC therapy is effective have not yet been reported. The investigators conducted a randomized clinical trial, extracted hair follicles from the human occipital area, prepared an HF-MSC suspension and locally injected it into the forehead hair loss area. Through follow-up observations, this study aimed to evaluate the safety and effectiveness of autologous hair follicle mesenchymal stem cell therapy in the treatment of AGA. The investigators expounded the possible effective population and stage.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Androgenic alopecia
* AGA classification include：The Norwood grade for male hair loss was II-V, and the Ludwig grade for female hair loss was I-III

Exclusion Criteria:

* (1) Using medications or supplements, including finasteride, dutasteride, ketoconazole, minoxidil or any other hormonal products, that can affect hair growth;
* (2) Patients with severe systemic diseases, immune diseases, endocrine diseases and nervous system diseases;
* (3) Patients with head skin infection, allergic disease and malignant tumor

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
hair diameters changed over time | 0 days, 1 month, 3 months, 6 months, and 9 months
  hair diameters changed over time

CONTACTS AND LOCATIONS:
Overall Officials: Zhiqi Hu, phD, Study Chair — southern hosptal
Locations (1):
- Department of Plastic and Aesthetic Surgery, Nanfang Hospital Southern 8 Medical University, Guangzhou, Guangdong, China